CLINICAL TRIAL: NCT04578522
Title: Correlation Between the Severity of Coronary Artery Disease and Peripheral Arterial Stiffness in Patients With Premature Coronary Heart Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Dongying Zhang, Clinical Professor, Chongqing Medical University
Other Study IDs: 2020-09-29
Record Dates: First submitted 2020-10-02; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Premature Coronary Heart Disease
Keywords: Premature coronary heart disease; Degree of coronary stenosis; arterial stiffness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Premature coronary heart disease (CHD) refers to the onset of myocardial infarction in men < 55 years old, women < 65 years old. At present, researches on early-onset coronary heart disease mostly focus on its risk factors and clinical characteristics, but there is no relevant research on the relationship between early-onset myocardial infarction and atherosclerosis.

DETAILED DESCRIPTION:
Premature coronary heart disease is defined as the first onset of male < 55 years old, female < 65 years old, confirmed by clinical examination. A number of studies have found that smokers have a significantly increased risk of acute myocardial infarction, and suggest that continued smoking is still an independent predictor of mace. These findings suggest that smoking is significantly associated with early-onset coronary heart disease. A number of studies have found that smoking can increase peripheral arterial stiffness. At present, there is no study on peripheral arterial stiffness in patients with early-onset myocardial infarction, so we suspect that peripheral arterial stiffness in patients with early-onset myocardial infarction is significantly increased

ELIGIBILITY:
Inclusion Criteria:

* The onset of coronary heart disease (including acute coronary syndrome and stable angina pectoris) was less than 55 years old in men and 65 years in women

Exclusion Criteria:

* Non coronary heart disease leading to chest pain (myocarditis, pericarditis, pulmonary embolism, aortic dissection, unstable angina pectoris) definite infection tumor liver and kidney insufficiency autoimmune disease acromegaly hyperthyroidism and subclinical hyperthyroidism secondary hypertension, etc.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with primary coronary heart disease were male < 55 years old and female < 65 years old
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-09-29 (Estimated); Primary Completion 2021-09-29 (Estimated); Study Completion 2021-09-29 (Estimated)

PRIMARY OUTCOMES:
Arterial stiffness | On admission
  The arterial stiffness of HFpEF patients, for exampleambulatory arterial stiffness indexbrachial ankle pulse wave velocity, ardioankle vascular index and so on.
Degree of coronary stenosis | On admission
  Degree of coronary stenosis indicated by coronary angiography

CONTACTS AND LOCATIONS:
Overall Officials: Dongying Zhang, doctor, Study Director — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, China